CLINICAL TRIAL: NCT03742804
Title: Pilot Phase 2 Study of Intratumoral G100 in Patients With Cutaneous T Cell Lymphoma
Brief Title: Study Of Intratumoral G100 In Cutaneous T Cell Lymphoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study sponsor sold and the new company would not support the study.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000021483
Record Dates: First submitted 2018-11-13; First posted 2018-11-15 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Lymphoma, T-Cell, Cutaneous
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- G100 injections (Experimental): All patients will receive 6 intratumoral G100 injections alone over 5 weeks. There will be a 4-week break for restaging. Patients will receive another 6 doses of G100 with either topical nitrogen mustard for 2 days before each dose or local radiotherapy (2 Gy daily x 2 days) prior to G100 to the injected lesion to assess the response to combination therapy. After the first 4 doses, nitrogen mustard is optional and can be omitted at the discretion of the investigator.
  Interventions: Biological: Intratumoral G100

INTERVENTIONS:
Biological: Intratumoral G100 — G100 agent is a potent Toll-like receptor (TLR)4 agonist. G100 is composed of glucopyranosyl lipid A (GLA) formulated in a stable emulsion (SE). GLA is a fully synthetic TLR4 agonist that is a potent stimulator of innate immune responses.

SUMMARY:
The overall goal of this study is to evaluate the safety and immunogenicity of repeat-dose intratumoral G100 administration in patients with Cutaneous T Cell Lymphoma (CTCL) alone (Part 1) and following standard local radiation therapy or topical nitrogen mustard application (Part 2). Plaque, patch, or tumor lesions of CTCL may be injected. Disease will be assessed in all sites, including skin, nodes, and blood.

DETAILED DESCRIPTION:
This is a pilot, Phase II study of intratumoral or intralesional injection of G100 alone (Part 1) and in conjunction with topical nitrogen mustard (HN2) or radiotherapy (Part 2) in patients with CTCL to generate anti-tumor immune responses. To confirm the safety of the injections in this population, enrollment of the first four patients will be staggered by at least 21 days each. If there are no grade 3 adverse events following the first 4 injections in the first 3 patients, then subsequent patients can be enrolled without restriction to timing.

Part 1: All patients will receive 6 intratumoral G100 injections alone over 5 weeks (first dose on Day 0, second on Day 5-7, and then weekly thereafter; up to Week 5) to assess the response to G100 alone. Response in target lesions will be measured by CAILS and abscopal effect will be measured by Modified Severity Weighted Assessment Tool (MSWAT). If applicable, peripheral blood flow cytometry will be used to assess response of circulating tumor cells.

There will be a 4-week break for restaging.

Part 2: Patients will receive another 6 doses of G100 with either topical nitrogen mustard for 2 days or local radiotherapy (2 Gy daily x 2 days) prior to G100 to the injected lesion to assess the response to combination therapy. After the first 4 doses, nitrogen mustard is optional and can be omitted at the discretion of the investigator. Response in target lesions will be measured by Composite assessment of index lesion severity (CAILS) and abscopal effect will be measured by MSWAT. If applicable, peripheral blood flow cytometry will be used to assess response of circulating tumor cells.

* Dose regimen interruption in a single patient may be made by the clinical investigator if it is deemed in the best interest of patient safety.
* Tumor imaging will be performed during the screening visit (baseline) in patients with blood involvement, palpable nodes, or tumor stage disease (scans done within 4 weeks of study entry are admissible), and in patients with clinically suspicious positive scans (nodes felt to be involved, standardized uptake value (SUV) 4 or greater on positron emission tomography (PET), imaging will be repeated at the completion of 6 weeks of dosing
* Circulating Sezary cells will be followed if present at baseline. Quantitation of Sezary cells will be done by flow cytometry using appropriate markers.
* Pre- and post-treatment tumor biopsies will be obtained for histologic review and exploratory immune analyses, including cell phenotype and genomic analyses of T cells. On-treatment biopsies will be performed at Week 3 of both Parts 1 and 2 of the study. Peripheral blood will be drawn for immune assays and other biomarker tests at time points listed in the Schedule of Events and Study Procedures.

Primary Objective

* To evaluate the safety and to observe clinical responses (by MSWAT and CAILS) with intratumoral G100 alone and with G100 in combination with agents to induce apoptosis (local radiotherapy or topical nitrogen mustard) in patients with CTCL.

Secondary Objectives

* To assess abscopal tumor responses in non-treated, distal tumor sites by MSWAT and CAILS tools.
* To evaluate pre-and post-regimen tumor tissue and blood for exploratory biomarkers of immunologic and tumor response.

ELIGIBILITY:
Inclusion Criteria:

1. Cutaneous T-cell lymphoma with persistent, relapsed or refractory disease following at least two prior therapies including at least one systemic therapy. Patients with aggressively progressing disease as per the investigator's assessment are not eligible.
2. Skin lesions accessible for intratumoral injection and at least one additional site of disease outside the radiation field for assessment of distal (abscopal) response.
3. ≥ 18 years of age.
4. Life expectancy of ≥ 6 months per the investigator.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Electrocardiogram (ECG) without evidence of clinically significant ischemia or arrhythmia
7. If female of childbearing potential (FCBP), willing to undergo pregnancy testing and agrees to use two methods of birth control or is considered highly unlikely to conceive during the dosing period and for three months after last study treatment.
8. If male and sexually active with a FCBP, must agree to use effective contraception such as latex condom or is sterile (e.g. following a surgical procedure) during the dosing period and for three months after last study treatment.

Exclusion Criteria:

1. Cancer therapies, including chemotherapy, radiation (non-study regimen related), within 4 weeks prior to the first scheduled G100 dose; histone deacetylase (HDAC) inhibitors and retinoids or interferon (IFN) or methotrexate or extracorporeal photopheresis (ECP) within 2 weeks
2. Investigational therapy within 4 weeks prior to G100 dosing
3. Inadequate organ function including:

   1. Marrow: Peripheral blood leukocyte count (WBC) < 3000/(cubic millimeter)mm3, absolute neutrophil count ≤ 1000/mm3, platelets < 100,000/mm3, or hemoglobin < 10 grams per deciliter (gm/dL).
   2. Hepatic: alanine aminotransferase (ALT), and aspartate aminotransferase (AST)> 2.5 x upper limit of normal (ULN), total serum bilirubin > 1.5 x ULN (patients withGilbert's Disease may be included if their total bilirubin is ≤3.0 (milligram) mg/dL)
   3. Renal: Serum creatinine ≤2 mg/dL
4. Significant immunosuppression from:

   1. Concurrent, recent (≤ 4 weeks ago) or anticipated treatment with systemic corticosteroids greater than a maintenance dose for adrenal insufficiency (10 mg daily)
   2. Other immunosuppressive medications (e.g.,methotrexate, cyclosporine, azathioprine)
5. Pregnant or nursing
6. Myocardial infarction within 6 months of study initiation, active cardiac ischemia or New YorkHeart Association (NYHA) Grade III or IV heart failure
7. History of other cancer within 2 years (except non-melanoma cutaneous malignancies, treated prostate cancer and cervical carcinoma in situ). Chronic lymphocytic leukemia (CLL) or low grade B-cell lymphoma will be considered on a case-by-case basis.
8. Recent (< 1 week ago) clinically significant infection or active tuberculosis or evidence of active hepatitis B, hepatitis C or human immunodeficiency virus (HIV) infection.
9. Central nervous system involvement with lymphoma, including parenchymal and leptomeningeal disease.
10. Significant autoimmune disease with the exception of alopecia, vitiligo, hypothyroidism or other conditions that have never been clinically active or were transient and have completely resolved and require no ongoing therapy.
11. Psychiatric, other medical illness or other condition that in the opinion of the principal investigator prevents compliance with study procedures or ability to provide valid informed consent.
12. History of significant adverse or allergic reaction to any component of G100 trial regimens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Clinical response will be assessed with the modified Severity Weighted Assessment Tool | From baseline through follow-up, up to 12 months.
  Clinical response will be assessed with the modified Severity Weighted Assessment Tool [mSWAT].
Clinical response will be assessed by the composite assessment of index lesion severity | From baseline through follow-up, up to 12 months.
  Clinical response will be assessed by the composite assessment of index lesion severity [CAILS])

SECONDARY OUTCOMES:
Abscopal tumor response will be assessed with the modified Severity Weighted Assessment Tool | From baseline through follow-up, up to 12 months.
  Tumor response will be assessed with the modified Severity Weighted Assessment Tool [mSWAT].
Abscopal tumor response will be assessed by the composite assessment of index lesion severity | From baseline through follow-up, up to 12 months.
  Tumor response will be assessed by the composite assessment of index lesion severity [CAILS]).

CONTACTS AND LOCATIONS:
Overall Officials: Francine Foss, MD, Principal Investigator — Yale University